CLINICAL TRIAL: NCT03138447
Title: A Digital Health Tool for Insulin Titration (DHIT) for Individuals With Type 2 Diabetes: A Prospective Outcomes Study With a Retrospective Control Group.
Brief Title: A Digital Health Tool for Insulin Titration (DHIT) Individuals With Type 2 Diabetes: A Prospective Outcomes Study With a Retrospective Control Group
Acronym: DHIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amalgam Rx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IS001
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: insulin; basal; titration; digital health
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: The design of this protocol involves a prospective and retrospective cohort. The prospective cohort includes 30 participants. In the retrospective chart review, participants will be matched to the prospective group for age, gender, and baseline A1C. (For this study, the use of the word 'matched' means that the retrospective patient charts will be matched as close as possible from available patient data within the Bay West Endocrinology medical record database and may not always be an exact match to the prospective group for age, gender, and baseline A1c.) The chart review will thus be conducted after the last subject is enrolled in the prospective arm of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Prospective Cohort (Experimental)
  Interventions: Device: Basal Insulin Titration Application
- Retrospective Cohort (No Intervention)

INTERVENTIONS:
Device: Basal Insulin Titration Application — Healthcare Providers ("HCP") and the principal investigator ("PI") will use an HCP portal to initiate a basal insulin titration algorithm. HCPs can customize the titration algorithm for every participant. Once a participant is prescribed an algorithm, they can download a mobile app on their phone with their HCPs corresponding titration plan. The app will prompt participants to enter their fasting glucose daily. Based on their fasting glucose and their HCPs titration plan, the application will display the participants daily basal insulin dose.
  Arms: Prospective Cohort

SUMMARY:
The digital health tool is an application ("app") available on iOS and Android enabled mobile phones. Health Care Providers ("HCPs") configure algorithms which can be tailored to individual patient's needs and then prescribe the app to support optimal basal insulin titration and dosing. In this study, participants will be recruited from a medical practice in which an HCP has prescribed a once-daily basal insulin. Participants will be trained on the use of the app utilizing their own mobile phone. During training, a brief self-assessment survey will be administered. After 90 days of usage, a telephone survey will be conducted. The baseline A1C results and the end of study A1C results will be collected from the patients' routine clinical care records. Data from the retrospective control group will be collected from a chart review of the same practice.

ELIGIBILITY:
Inclusion Criteria:

- Prospective cohort: The participants will be patients with type 2 diabetes mellitus who are not at goal on their current dose of prescribed basal insulin (e.g. Lantus, Toujeo, Levemir, Tresiba, or Basaglar). Participants shall be age 21 or older, prescribed basal insulin within the past 18 months, own a compatible mobile phone, able to receive/make calls and read messages on their phone. There is no predefined gender or ethnic group. Participants should be generally healthy and not expected to be hospitalized for surgery or other medical care during the study period.

- Retrospective cohort: This will be a chart review. Participants will be matched to the prospective cohort for age, gender and baseline A1C. Patients should have been prescribed one of the basal insulins above.

Exclusion Criteria:

- Prospective cohort: Participants with stage 4 or 5 kidney disease, active malignancies, variable glucocorticoid doses during the study period, severe visual impairment, or dementia will be excluded. Also, participants prescribed rapid-acting or premixed insulins (any insulin not on the above list) will be excluded.

- Retrospective cohort: Same as above.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Basal Insulin Dose | 90 days
  Change in basal insulin dose from entry into study to completion of study.

SECONDARY OUTCOMES:
Change in Fasting Glucose | 90 days
  Change in the average fasting blood glucose in the final week of the study as compared to the first week of the study.
Fasting Glucose in Target | 90 days
  Proportion of participants whose fasting blood glucose is in the ADA target range by the end of the 90 day study period.
Titration Adherence | 90 days
  Proportion of participants who adhered to their basal insulin dose adjustments according to their algorithm.
Change in A1C | 90 days
  Change in hemoglobin A1C measure at the completion of the study as compared to baseline.
Change in Diabetes Distress | 90 days
  Change in measures of diabetes distress at the completion of the study as compared to baseline.
Participant Satisfaction | 90 days
  Demonstration of satisfaction with the app at the completion of the study.
Office Contacts | 90 days
  Reduction in number of HCP contacts (live office visits and phone calls) regarding insulin management during 90 day period.

CONTACTS AND LOCATIONS:
Locations (1):
- MODEL Clinical Research, Towson, Maryland, United States

IPD SHARING:
Plan to Share IPD: No